CLINICAL TRIAL: NCT00403260
Title: A Phase III Comparative, Open-label, Randomised, Multi-centre Study to Assess the Efficacy of Pyronaridine Artesunate (180:60mg) Versus Mefloquine (250mg) Plus Artesunate (100mg) in Children & Adult Patients With Acute Falciparum Malaria
Brief Title: Pyronaridine - Artesunate (3:1) Versus Mefloquine Plus Artesunate in Plasmodium Falciparum Malaria Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-004-06
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Falciparum Malaria
Keywords: malaria; antimalarial; P falciparum; pyronaridine; artesunate; artemisinin based combination therapy (ACT); pyronaridine artesunate (Pyramax)
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; Mefloquine; Artesunate

ARMS (2):
- Pyronaridine - artesunate (Experimental): Oral pyronaridine artesunate (180:60mg tablets) once a day for 3 consecutive days (Day 0, 1, and 2). Posology based on body weight ranges.
  Interventions: Drug: Pyronaridine - artesunate
- Mefloquine plus artesunate (Active Comparator): Mefloquine (250mg tablets) plus artesunate (100mg tablets) once a day for 3 consecutive days (Day 0, 1, and 2). Posology based on body weight ranges.
  Interventions: Drug: Mefloquine plus artesunate

INTERVENTIONS:
Drug: Pyronaridine - artesunate — once a day for 3 days
  Other Names: Pyramax
  Arms: Pyronaridine - artesunate
Drug: Mefloquine plus artesunate — once a day for 3 days
  Arms: Mefloquine plus artesunate

SUMMARY:
The primary objective of this phase III clinical study is to compare the efficacy and safety of the fixed combination of pyronaridine artesunate (Pyramax®, PA) with that of the combination of mefloquine plus artesunate (MQ + AS) in children and adults with uncomplicated P falciparum malaria in South East Asia, India and Africa.

DETAILED DESCRIPTION:
This is a multi-centre, comparative, randomised, open-label, parallel-group, non-inferiority study comparing the efficacy and safety of a fixed combination of PA to a loose combination of MQ + AS for patients with acute, symptomatic, uncomplicated P. falciparum malaria. The study population will include 1271 patients, comprising male and female children (≥20 kg body weight) and adults, recruited from study sites in South East Asia, India and Africa. Patients will be randomised in a 2:1 ratio to receive either oral PA (180:60mg tablets) or MQ (250mg tablets) plus AS (100mg tablets) once a day for 3 consecutive days (Days 0, 1, and 2). The study drug will be administered by a Third-Party Investigator unblinded to the study treatment, while the Investigator remains blinded.

Patients will be confined to the to the study facility for ≥4 days (Days 0, 1, 2, and 3) and remain near the study site for ≥7 days, or once fever and parasite clearance has been confirmed for ≥24 hours - whichever occurs later.

The primary efficacy end point for the study is the proportion of patients with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28. Scheduled follow-up visits will continue until completion of the study at Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

The primary efficacy end point for the study is the proportion of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28 (defined as the absence of parasitaemia without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure). Scheduled follow-up visits will continue until completion of the study at Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 3 and 60 years, inclusive.
* Body weight between 20 kg and 90 kg with no clinical evidence of severe malnutrition.
* Presence of acute uncomplicated P. falciparum mono-infection confirmed by:

  1. Fever, as defined by axillary/tympanic temperature ≥37.5°C or oral/rectal temperature ≥38°C, or documented history of fever in the previous 24 hours and,
  2. Positive microscopy of P. falciparum with parasite density between 1,000 and 100,000 asexual parasite count/µl of blood
* Written informed consent provided by patient and/or parent/guardian/spouse.
* Ability to swallow oral medication.

Exclusion Criteria:

* Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organization Criteria 2000.
* Mixed Plasmodium infection.
* Severe vomiting or severe diarrhoea.
* Known history or evidence of clinically significant disorders.
* Presence of significant anaemia, as defined by Hb <8 g/dL.
* Presence of febrile conditions caused by diseases other than malaria.
* Known history of hypersensitivity, allergic or adverse reactions to pyronaridine, mefloquine or artesunate or other artemisinins.
* Use of any other antimalarial agent within 2 weeks prior to start of the study as evidenced by positive urine test.
* Female patients of child-bearing potential must be neither pregnant (as demonstrated by a negative pregnancy test) nor lactating, and must be willing to take measures to not become pregnant during the study period.
* Presence of significant renal or hepatic impairment.
* Receipt of an investigational drug within the past 4 weeks.
* Known active Hepatitis A IgM, Hepatitis B surface antigen or Hepatitis C antibody.
* Known seropositive HIV antibody.
* Previous participation in any clinical study with PA.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1271 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Borghini-Fuhrer, PhD, Study Director — Medicines for Malaria Venture
Locations (9):
- RAOTAP2/Centre Muraz, Bobo-Dioulasso, Houet Province, Burkina Faso
- Pailin Referral Hospital, Pailin, Pailin, Cambodia
- Institut Pasteur, Abidjan, Côte d’Ivoire
- Wentlock District Hospital, Mangalore, India
- Bagamoyo Research and Training Centre of Ifakara Health Institute, Bagamoyo, Tanzania
- Thailand (2):
  - MaeLamad District Hospital, Mae Ramat, Changwat Tak
  - MaeSod General Hospital, Mae Sot, Changwat Tak
- Vietnam (2):
  - NIMPE, Hanoi, Commune Xy
  - Choray Hospital, Dak O, Ho Chi Minh City

REFERENCES:
- [Result] Rueangweerayut R, Phyo AP, Uthaisin C, Poravuth Y, Binh TQ, Tinto H, Penali LK, Valecha N, Tien NT, Abdulla S, Borghini-Fuhrer I, Duparc S, Shin CS, Fleckenstein L; Pyronaridine-Artesunate Study Team. Pyronaridine-artesunate versus mefloquine plus artesunate for malaria. N Engl J Med. 2012 Apr 5;366(14):1298-309. doi: 10.1056/NEJMoa1007125. PMID 22475593
- [Derived] Ayyoub A, Methaneethorn J, Ramharter M, Djimde AA, Tekete M, Duparc S, Borghini-Fuhrer I, Shin JS, Fleckenstein L. Population Pharmacokinetics of Pyronaridine in Pediatric Malaria Patients. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1450-8. doi: 10.1128/AAC.02004-15. PMID 26666916
- [Derived] Duparc S, Borghini-Fuhrer I, Craft CJ, Arbe-Barnes S, Miller RM, Shin CS, Fleckenstein L. Safety and efficacy of pyronaridine-artesunate in uncomplicated acute malaria: an integrated analysis of individual patient data from six randomized clinical trials. Malar J. 2013 Feb 21;12:70. doi: 10.1186/1475-2875-12-70. PMID 23433102

RESULTS

PARTICIPANT FLOW:
Groups:
- Pyronaridine - Artesunate: Pyronaridine - artesunate (180:60mg) once a day for 3 days. Posology was based on body weight ranges.
- Mefloquine Plus Artesunate: Mefloquine (250mg) plus artesunate (100mg) once a day for 3 days. Posology was based on body weight ranges.
Period: Overall Study
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Started | 848 (Patients randomized and treated.) | 423 (Patients randomized and treated.)
Completed | 723 | 357
Not Completed | 125 | 66
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 49 | 25
Not completed — Re-appearance of P. falciparum | 34 | 25
Not completed — P. vivax infection | 26 | 4
Not completed — Mixed infection with P. vivax | 2 | 0
Not completed — Mixed infection with P. falciparum | 1 | 0
Not completed — P. vivax infection at screening | 1 | 0
Not completed — P. ovale infection | 1 | 0
Not completed — Gametocyte re-appearance | 1 | 1
Not completed — Withdrawn from study accidentally | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population, consisted of all randomized subjects who received any amount of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate | Total
Number analyzed (Participants) | 848 | 423 | 1271
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (11.67) | 25.4 (12.54) | 25.1 (11.96)
Age, Continuous [Median (Full Range); unit: years] | 23 [4 to 60] | 23.0 [5 to 59] | 23.0 [4 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214 | 93 | 307
  Male | 634 | 330 | 964
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 689 | 344 | 1033
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 159 | 79 | 238
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 108 | 55 | 163
  Burkina Faso | 83 | 39 | 122
  Cambodia | 140 | 71 | 211
  Tanzania | 25 | 13 | 38
  Côte D'Ivoire | 51 | 27 | 78
  Thailand | 402 | 198 | 600
  India | 39 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With PCR-corrected Adequate Clinical and Parasitological Response (ACPR) on Day 28
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28, defined as absence of parasitaemia on Day 28 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure.
Time Frame: Day 28
Population: Efficacy evaluable population subjects completed a full course of study med., did not miss a dose, did not use a concomitant med. that may have interfered with the treatment outcome up to D14, did not have a concomitant disease which may have interfered with the classification of the treatment outcome, and did not have major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 749 | 367
percentage of subjects | 99.2 [98.3 to 99.7] | 98.1 [96.1 to 99.2]
Statistical Analysis 1: Comparison: Pyronaridine - Artesunate vs Mefloquine Plus Artesunate; Null hypothesis: The PCR-corrected ACPR response rate at Day 28 for the PA group is inferior to the PCR-corrected ACPR response rate at Day 28 for the comparator group (MQ + AS) by more than 5%. Was tested versus the alternative: Alternative hypothesis: the PCR-corrected ACPR response rate at Day 28 for the PA group is not inferior to the PCR-corrected ACPR response rate at Day 28 for the comparator group (MQ + AS) by more than -5%; Test type: Non-Inferiority or Equivalence — The primary efficacy analysis tested the non-inferiority of the PA group compared to the comparator group with regard to the PCR-corrected ACPR response rate at Day 28 using the 2-sided 95% confidence interval (CI) (Newcombe-Wilson score method without continuity correction). Non-inferiority of PA to MQ + AS was concluded if the lower limit of the CI for the difference was >-5%; p = 0.106, Chi-squared — If non-inferiority of PA was demonstrated, the p-value associated with a superiority test is calculated based on a 2-sided Chi-square test. If the calculated p-value is <5%, then the superiority of PA compared to MQ+AS was statistically demonstrated; ACPR percent difference = 1.1, 95% CI 2-sided [-0.2 to 3.1]

2. Secondary Outcome: PCR-corrected ACPR on Day 14
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 14, defined as absence of parasitaemia on Day 14 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Day 14
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 749 | 367
percentage of subjects | 99.9 [99.3 to 100.0] | 99.5 [98.0 to 99.9]

3. Secondary Outcome: Crude ACPR on Days 14 and 28
Description: Percentage of subjects with adequate clinical and parasitological response (ACPR) on Days 14 and 28, without correction by PCR, defined as absence of parasitaemia on Days 14 and 28 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Days 14 and 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 749 | 367
percentage of subjects
  Cure rate (%) on Day 14 | 99.9 [99.3 to 100.0] | 99.5 [98.0 to 99.9]
  Cure rate (%) on Day 28 | 98.7 [97.6 to 99.4] | 96.7 [94.4 to 98.3]

4. Secondary Outcome: Parasite Clearance Time
Description: Parasite clearance time was defined as the time from first dosing to time of first blood draw with parasite clearance. Parasite clearance was defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart.
Time Frame: Thick blood films were examined every 8 hours until ≥72 hours or until 2 consecutive negative readings occurred 7 to 25 hours apart, and on Days 3, 7, 14, 21, 28, 35, and 42 (or any other day if the subject returned).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 749 | 367
hours | 31.7 [31.4 to 31.8] | 32.0 [31.8 to 36.8]

5. Secondary Outcome: Fever Clearance Time
Description: Fever clearance time was defined as the time from first dosing to first normal reading of temperature (<37.5°C taken axillary or tympanic; <38°C taken oral or rectal) for 2 consecutive normal temperature readings taken between 7 and 25 hours apart.
Time Frame: Every 8 hours over ≥72 hours following first study drug administration or temperature normalisation for ≥2 readings between 7 and 25 hours apart, then at each visit.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 627 | 313
hours | 15.9 [15.7 to 16.0] | 16.0 [15.7 to 16.0]

6. Secondary Outcome: Parasite Clearance at Day 1, 2 and 3
Description: Parasite clearance time was defined as the time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance was defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 749 | 367
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 38.5 [35.1 to 42.0] | 31.6 [27.1 to 36.6]
  Clearance rate (%) at Day 2 (48h after first dose) | 83.8 [81.1 to 86.4] | 79.8 [75.6 to 83.8]
  Clearance rate (%) at Day 3 (48h after first dose) | 91.5 [89.3 to 93.3] | 90.5 [87.2 to 93.2]

7. Secondary Outcome: Fever Clearance at Day 1, 2 and 3
Description: Fever clearance time was defined as the time for at least 2 consecutive normal body temperature measurements (<37.5°C axillary/tympanic or <38.0°C oral/rectal) to be obtained within an interval of 7 to 25 hours post-dosing.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 627 | 313
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 78.5 [75.2 to 81.6] | 78.9 [74.2 to 83.2]
  Clearance rate (%) at Day 2 (48h after first dose) | 95.9 [94.1 to 97.2] | 96.2 [93.6 to 99.9]
  Clearance rate (%) at Day 3 (72h after first dose) | 99.2 [98.2 to 99.7] | 98.4 [96.5 to 99.4]

8. Secondary Outcome: Adverse Events and Clinically Significant Laboratory Results
Description: Cases and severity of adverse events and of clinically significant laboratory results, ECG, vital signs or physical examination abnormalities
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Population: The safety population consisted of all randomised subjects who received any amount of study medication; subjects were analysed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
Number analyzed (Participants) | 848 | 423
Participants
  Nr subj. with ≥1 AE | 389 | 190
  Nr subj. with ≥1 treatment-related AE | 153 | 94
  Nr subj. with ≥1 SAE | 6 | 3
  Nr subj. with ≥1 treatment-related SAE | 0 | 2
  Nr subj. with ≥1 severe or life threatenining AE | 24 | 23
  Nr subj. with ≥1 AE leading to death | 0 | 0
  Nr subj with ≥1 AE leading to drug discontinuation | 5 | 4
  Nr subj. with ≥1 AE leading to study withdrawal | 5 | 4

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Description: An AE was defined as any unfavorable and unintended sign, symptom, syndrome, or illness that developed or worsened during the period of observation in the clinical study.
Groups:
- Pyronaridine - Artesunate: Pyronaridine artesunate (180:60mg)
  Pyronaridine artesunate: once a day for 3 days
- Mefloquine Plus Artesunate: Mefloquine (250mg) plus artesunate (100mg)
  Mefloquine plus artesunate: once a day for 3 days
Arm/Group | Pyronaridine - Artesunate | Mefloquine Plus Artesunate
All-Cause Mortality (participants affected / at risk) | 0/848 | 0/423
Serious Adverse Events (participants affected / at risk) | 6/848 | 3/423
Other Adverse Events (participants affected / at risk) | 389/848 | 190/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine - Artesunate (N=848) | Mefloquine Plus Artesunate (N=423)
Cholera (Infections and infestations) | 1 (1) | 0 (0) — Cholera Inaba
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Transient auto immune hemolytic anemia
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1) — Tonic clonic seizure. Treatment-related SAE.
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) — Seizure. Treatment related SAE.
Cerebral malaria (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine - Artesunate (N=848) | Mefloquine Plus Artesunate (N=423)
Myalgia (Musculoskeletal and connective tissue disorders) | 53 (60) | 19 (20)
Dizziness (Nervous system disorders) | 26 (26) | 28 (29)
Headache (Nervous system disorders) | 101 (120) | 44 (48)
Anorexia (Metabolism and nutrition disorders) | 39 (41) | 13 (13)
Anaemia (Blood and lymphatic system disorders) | 31 (31) | 17 (17)
Basophilia (Blood and lymphatic system disorders) | 8 (8) | 9 (9)
Eosinophilia (Blood and lymphatic system disorders) | 20 (20) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 14 (14) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 9 (9)
Nausea (Gastrointestinal disorders) | 9 (9) | 8 (8)
Vomiting (Gastrointestinal disorders) | 18 (18) | 9 (9)
Fatigue (General disorders) | 16 (18) | 6 (6)
Pyrexia (General disorders) | 12 (12) | 4 (4)
Bronchitis (Infections and infestations) | 15 (15) | 6 (6)
Nasopharyngitis (Infections and infestations) | 21 (21) | 11 (11)
Alanine aminotransferase increased (Investigations) | 21 (21) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (19) | 1 (1)
Blood creatinine phosphokinase increased (Investigations) | 12 (12) | 4 (4)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 5 (5)
Eosinophil count increased (Investigations) | 9 (9) | 6 (6)
Haemoglobin decreased (Investigations) | 21 (21) | 7 (7)
Platelet count increased (Investigations) | 10 (10) | 3 (3)
Transaminases increased (Investigations) | 18 (18) | 3 (3)
Insomnia (Psychiatric disorders) | 13 (13) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (33) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No